CLINICAL TRIAL: NCT06536634
Title: Effects and Mechanisms of Sensory Afferent Electrostimulation on Upper Limb Function in Patients With Hemiparesis
Acronym: SAES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-00982
Record Dates: First submitted 2024-07-10; First posted 2024-08-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hemiparesis; Unilateral Cerebral Palsy
Keywords: Sensory afferent electrostimulation; MRI; TMS; Motor function; Sensory function; Sensor
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Intervention Model Description: A randomized controlled Bayesian phase II trial with a follow-up examination after 12 weeks mwas designed. The study participants will be recruited via the University Children's Hospital Bern and the Swiss Cerebral Palsy Registry.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAES (Experimental): Treatment group (SAES)
  Interventions: Sensory afferent electrical stimulation (SAES)
  Interventions: Other: SAES
- Control group (Other): The control intervention (treatment as usual, TAU) consists of the prescribed conventional occupational therapy and/or physiotherapy.
  Interventions: Other: TAU

INTERVENTIONS:
Other: SAES — The experimental intervention consists of SAES with a glove or adhesive electrodes at 20Hz, 300µs, intensity between 2-10mA, during 30 minutes per day, 5x/week, for 5 weeks, combined with conventional occupation therapy. The subsequent therapy sessions will take place at home, with in-between telephone checks.
  Arms: SAES
Other: TAU — Treatment as usual
  Arms: Control group

SUMMARY:
The goal for this project is to investigate the effects of a 5-week SAES therapy in addition to conventional therapy on both behavioural (sensory and motor) and neurological measures and the underlying mechanisms of treatment response.

The goal of this project to investigate the effects of a 5-week SAES therapy in addition to conventional therapy.

The aim is to investigate whether SAES is more effective than conventional therapy alone in children with hemiparesis. The investigators will assess the efficacy of SAES using novel clinical assessment such as kinematic evaluations and modern neurophysiological measures, namely transcranial magnetic stimulation (TMS) and resting-state functional MRI (rs-fMRI).

It will be expected a benefit for children with hemiparesis after SAES training which may lead to improved bimanual and unimanual functions. Benefits have been reported in adults and in preliminary studies also in children.

Type of study: Randomised controlled clinical trial

Participants with hemiparesis will be included in the study. The study group will receive the SAES training with a glove or adhesive electrodes as a home-based training during 30 minutes per day, 5x/week, for 5 weeks, combined with conventional occupation therapy.

Researchers will compare the SAES group with a group of patients with comparable conditions who receive the prescribed conventional occupational therapy and/or physiotherapy (treatment as usual, TAU)

DETAILED DESCRIPTION:
Children with hemiparesis present with sensory and motor deficits, which negatively affect quality of life and decrease participation in everyday life. To date, no treatment is yet effective to decrease these impairments. A recent systematic review confirms that unimanual and bimanual trainings effectively improve upper limb function in children with hemiparesis. However, it is still challenging to find the best individual training method for children with hemiparesis, as there is much variability in treatment response.

In the present study, the effects and mechanisms of non-invasive electrostimulation of the hand, called Sensory Afferent Electrostimulation (SAES) will be investigated. SAES triggers action potentials in afferent nerve fibres leading to increased sensory afferent input in the sensorimotor regions of the brain. Through this, SAES can enhance excitability of the motor cortex and of upper limb performance. While proven effective in adults after stroke, SAES is safe with promising positive results in a very small study in children with hemiparesis. However, the investigation of efficacy of SAES on sensory and motor functions was so far neglected. Modern stimulation and imaging methods revealed that, whole-hand SAES induced increased strength of corticospinal projections and intracortical change (measured with transcranial magnetic stimulation), which may indicate long-term potentiation mechanisms. Furthermore, in a functional MRI study, SAES induced increased motor cortex activity. Hence, resting state fMRI will allow to understand the efficacy of SAES on the topographically connectivity of the motor and sensorimotor network at rest.

The experimental intervention consists of SAES with a glove or adhesive electrodes (e.g. Cefar Reha X2) at 20Hz, 300µs, intensity between 2-10mA, during 30 minutes per day, 5x/week, for 5 weeks, combined with conventional occupation therapy. The subsequent therapy sessions will take place at home, with in-between telephone checks.

The control intervention (treatment as usual, TAU) consists of the prescribed conventional occupational therapy and/or physiotherapy. The evaluation of the UL sensory and motor function will be conducted at the University Children's Hospital in Bern by blind assessors, expert in the clinical measures, and will take place before and after each intervention period and at 12-weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral cerebral palsy/hemiparesis, following unilateral brain lesion, e.g. perinatal/childhood stroke (acquired prior to the age of 16 years)
* consistent and stable limitation of hand functions
* chronic state (time since lesion >2 years)
* aged 6-18 years
* parental informed consent if <14 years, informed consent of the patient if >14 years

Exclusion criteria:

* psychiatric disease that prevents the participant form informed participation and compliance in an adequate manner/setting
* Bilateral brain lesion
* Recent Botulinum toxin-injections injections (UL, < 6 months)
* Hand surgery on paretic hand < 2 years
* Trauma to UL in the last year
* Medical conditions that prevent training of the UL
* Participation in other afferent stimulation studies
* Electrical stimulation therapy in the last 6 months
* Intensive training of the UL (therapy more than 1x/week, < 6 months)

If MRI and TMS is performed, additionally:

• MRI and TMS contradictions, such as

* implanted Metal devices (e.g. braces, implant)
* implanted shunt system
* in girls and women: pregnancy
* claustrophobia
* Active epilepsy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Bimanual hand function | 5 weeks (After the treatment)
  Will be measured with the Assisting Hand Assessment (AHA)

SECONDARY OUTCOMES:
Bimanual hand function | 2 assessments: baseline, follow up (12 weeks)
  Will be measured with the Assisting Hand Assessment (AHA)
Bimanual hand function in everyday life activities | 2 assessments: baseline, follow up (12 weeks)
  Will be measured with the Chedoke Arm and Hand Activity Inventory (CAHAI)
Spasticity | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Modified Ashworth scale)
Strength | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Dynamometer)
Sensitivity | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Semmes-Weinstein monofilaments)
Unimanual hand function | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Jebson-Taylor Hand function test)
Stereognosis | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Stereognosis test with Jamar toolkit)
Hand function during daily activities | 2 assessments: baseline, after the treatment (5 weeks)
  Will be assessed via questionnaires (CHEQ)
Mirror movements | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via clinical assessments (Woods and Teuber Scale)
Hand/wrist position | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  The Zancolli Wrist Classification categorizes the most commonly observed wrist and hand deformities of children with spastic CP and the relative contributions of intrinsic and extrinsic muscles to hand deformity and function.
Hand/Finger position | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  To measure the hand/finger position the House classification for the thumb in palm pattern will be assessed.
Upper limb kinematic activity | 2 assessments: baseline, after the treatment (5 weeks)
  Will be assessed with novel sensory measures in an instrumented apartment using DeepLabCut software
MRI - Neurophysiological outcomes | 2 assessments: baseline, after the treatment (5 weeks)
  Magnetic resonance imaging (MRI) of the brain will be conducted in a 3-T scanner, lasting approximately one hour (including preparation). Structural (T1-weighted and T2-weighted) and FLAIR imaging will be performed. Resting-state functional MRI (rs-fMRI) will be used to study the spontaneous fluctuations in blood oxygen level dependent (BOLD) signal.
  Arterial spin labelling will be performed to assess blood flow imbalance.
TMS - Neurophysiological outcomes | 2 assessments: baseline, after the treatment (5 weeks)
  Neuro-navigated TMS will be used at the Department for Neurosurgery at the University Hospital Bern. Neuro-navigated TMS allows a 3D brain reconstruction to topographically map the neurophysiological responses at the cortical and subcortical levels, using single-pulse (resting and active motor thresholds, motor evoked potential amplitudes and latencies and stimulus recruitment curves) and paired-pulse (intracortical interactions) protocols.
Quality of life of Children with hemiparesis | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via the Kidscreen-52 questionnaire, which was designed to address generic health related quality of life.
Quality of life of Children with hemiparesis regarding hand function | 3 assessments: baseline, after the treatment (5 weeks), follow up (12 weeks)
  Will be assessed via the Children's Hand-use Experience Questionnaire (CHEQ). It has been developed for children and adolescents with decreased function in one hand, to evaluate the experience of children and adolescents in using the affected hand in activities where usually two hands are needed.
Reported Pain | Daily during the treatment phase (duration of treatment phase 5 weeks)
  Will be assessed via a visual analogue scale regarding the experienced pain on the paretic hand before and after the electrical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Regula Everts, Prof. Dr., Study Chair — Insel Gruppe AG, University Hospital Bern; Grunt Sebastian, Prof. Dr., Principal Investigator — Insel Gruppe AG, University Hospital Bern; Nef Tobias, Prof. Dr., Study Chair — ARTORG; Wiest Roland, Prof. Dr., Study Chair — Insel Gruppe AG, University Hospital Bern; Seidel Kathleen, Prof. Dr., Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No